CLINICAL TRIAL: NCT05002686
Title: Safety and Efficacy of Sintilimab in Combination With Albumin-Paclitaxel/Oxaliplatin/Capecitabine and Radiotherapy Followed by D2 Surgical Resection in Patients With Advanced Gastric Cancer With Retroperitoneal Lymph Node Metastasis: A Multiple Center Single Arm Trial
Brief Title: Safety and Efficacy of Sintilimab in Combination With Chemoradiothrapy Followed by D2 Surgical Resection in Patients With Advanced Gastric Cancer With Retroperitoneal Lymph Node Metastasis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Chen Li, Chief physician, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dragon VIII
Record Dates: First submitted 2021-08-10; First posted 2021-08-12 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Gastric Cancer
Keywords: retroperitoneal lymph node metastasis; chemoradiotherapy; surgical resection
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; Capecitabine; Oxaliplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab+ Albumin-Paclitaxel+Oxaliplatin +capecitabine+radiothrerapy+D2 Surgical Resection (Experimental)
  Interventions: Drug: Sintilimab; Drug: Albumin-Paclitaxel; Drug: Capecitabine; Drug: Oxaliplatin; Radiation: Radiation; Procedure: Radical gastric cancer surgery

INTERVENTIONS:
Drug: Sintilimab — 200 mg Q3W on Day 1 by IV infusion
  Other Names: IBI308
Drug: Albumin-Paclitaxel — 200 mg/m^2 Q3W on Day 1 by IV infusion
Drug: Capecitabine — 1000 mg/m^2 orally according to Body Surface Area (BSA) BID Q3W on Days 1-14
Drug: Oxaliplatin — 130 mg/m^2 Q3W on Day 1 by IV infusion
Radiation: Radiation — Radiotherapy for gastric lesions and high-risk areas of retroperitoneal lymph node before sugery, 45Gy*25.
Procedure: Radical gastric cancer surgery — Radical gastric cancer surgery with D2 lymph node dissection

SUMMARY:
Gastric cancer with retroperitoneal lymph node metastasis was considered as unresectable, to improve these patients' prognosis, we designed systematic conversion therapy including immunotherapy and chemoradiotherapy. The purpose of this study is to estimate safety and efficacy of Sintilimab in combination with chemoradiothrapy followed by D2 surgical resection in patients with advanced gastric cancer with retroperitoneal lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Pathology confirmed Gastric/Gastricgastroesophageal junction adenocarcinoma;
* Radiolgical imging including CT,PET-CT or MRI diagnosed as retroperitoneal metastasis.
* Did not receive previous systemic treatment (chemotheray, radiotherapy or both) for advanced disease before.
* ECOG PS 0-2.
* Adequate organ and bone marrow functions and life expectancy ≥12 weeks.

Exclusion Criteria:

* Distant metastases except retroperitoneal metastasis (liver, lung, peitoneal metastasis...);
* HER2-positive status;
* Suspicious active bleeding or gastriointestineal obstruction phenomenon and Has difficulty in swallow tablets and food;
* Has received prior therapy with an anti-programmed death (PD)-1, anti-PD-L1, anti-PD L2 , anti-CD137,anti-CTLA-4 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
* Is currently participating in and receiving study therapy ,except those in the survival follow up period of an investigational agent study or non-interventional study .
* Received systemic treatment with corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 4 weeks of first dose. Inhaled or topical steroids ,adrenal replacement steroid doses and steroid of prevention allergic reaction of i.v. contrast agent are permitted in the absence of active autoimmune disease.
* Known acute or chronic active hepatitis B infection (positive HBsAg and HBV DNA ≥ 200 IU/mL or ≥ 10^3 copies/mL positive) infection or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA positive) infection.
* Women who are pregnant or nursing.
* Received a live vaccine within 4 weeks of the first dose of study medication or plan to receive live vaccine during study period.
* Active, known or suspected autoimmune disease or has a history of the disease within the last 2 years (subjects with vitiligo, psoriasis, alopecia or Grave's disease, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or type I diabetes mellitus only requiring insulin replacement, but not required systemic treatment in the last 2 years, are permitted to enroll) .
* Known primary immunodeficiency.
* Known active tuberculosis.
* Known history of allogeneic organ or allogeneic hemopoietic stem cell transplantation.
* Known>=grade 3 allergy or hypersensitivity to Albumin-paclitaxel oxaliplatin, capecitabine or any monoclonal antibodies.
* Human Immunodeficiency Virus (HIV) infection (HIV antibody positive).
* Poorly controlled arterial hypertension (SBP ≥ 160mmHg or DBP ≥ 100 mmHg) with standard treatment .
* Symptomatic congestive heart failure (New York Heart Association grade II-IV) or symptomatic, poorly controlled arrhythmia.
* Prior arterial thromboembolism event, including myocardial infarction, unstable angina, stroke and transient ischemic attack, within 6 months of enrollment.
* Active or poorly controlled severe infection.
* History of gastrointestinal perforation and /or fistula within 6 months before enrollment.
* Other acute or chronic diseases, mental illness, or abnormal laboratory test results that may lead to the following outcomes: increase the risk of participating in study or study drug administration, or interfere with the interpretation of the study results and considered by investigator as "NOT" eligible to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-07 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
1 year Progression Free Survival (PFS) | Approximately 3 years after the first participant is included

SECONDARY OUTCOMES:
R0 surgical resection percentage | Approximately 2 years after the first participant is included
Operative conversion percentage | Approximately 2 years after the first participant is included
Overall survival (OS) | Approximately 4 years after the first participant is included
Number of participants experiencing clinical and laboratory adverse events (AEs) | Approximately 4 years after the first participant is included
Percentage of pathologic complete response(pCR) | Approximately 2 years after the first participant is included

OTHER OUTCOMES:
Potential biomarker to predict prognosis | Approximately 4 years after the first participant is included
  PD-L1 CPS, EBV expression, Tumor Mutational Burden(TMB), MSI-H/dMMR

CONTACTS AND LOCATIONS:
Overall Officials: Chen Li, PhD, Principal Investigator — Ruijin hospital affiliatted to Shanghai Jiaotong University school of medicine
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China